CLINICAL TRIAL: NCT06459765
Title: Mi2000 Totally Implantable Cochlear Implant (Mi2000 TICI): Pivotal Study
Brief Title: Mi2000 Totally Implantable Cochlear Implant (Mi2000 TICI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-EL_CRD_2021_02
Record Dates: First submitted 2024-06-03; First posted 2024-06-14 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional Arm (Experimental): Implantation with Mi2000 TICI
  Interventions: Device: Mi2000 TICI

INTERVENTIONS:
Device: Mi2000 TICI — Cochlear Implantation

SUMMARY:
The goal of this clinical trial is to test the Mi2000 Totally Implantable Cochlear Implant in a population of candidates for a cochlear implant. The main question it aims to answer is, whether the device is able to improve speech perception compared to the pre-operative score.

Participants will undergo cochlear implantation and fitting, and will be asked to perform the following tests pre- and post-operatively:

* Word test in quiet
* Sentence test in noise
* Audiograms
* Health Utilities Index 2 and 3 (HUI2&3), a generic quality-of-life questionnaire
* Nijmengen Cochlear Implant Questionnaire (NCIQ), a disease specific quality-of life questionnaire
* Speech, Spatial and Qualities of Hearing Scale (SSQ12), a disease specific questionnaire
* Hearing Implant Sound Quality Index (HISQUI19), a sound quality questionnaire

DETAILED DESCRIPTION:
Cochlear implants (CI) provide a large majority of recipients with a significant degree of speech understanding. However, CI systems rely on external audio processors to function. This can have several disadvantages: for instance, the hardware is exposed to external trauma and to the effects of head movement and gravity. The device is also put at risk by humid, dusty, or dirty conditions as well as by physical activities that lead to water exposure such as swimming or sports in general (e.g. perspiration).

In addition, some patients are concerned with the cosmetic appearance of the external parts which are visible (more so than modern behind-the-ear hearing aids), something that may not be desirable to many potential candidates.

This clinical investigation aims to collect confirmatory data on the use of the Mi2000 Totally Implantable Cochlear Implant system used in combination with compatible devices.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of eighteen (18) years at time of enrolment
* Bilateral sensorineural hearing loss with no or limited benefit from a hearing aid (>70 dB HL PTA4)
* Post-lingual onset of deafness
* No or limited benefit from hearing aids for less than 10 years and an expected benefit from cochlear implantation
* A maximum score of 50% on a word test in the language of the test centre in the ear to be implanted in the best aided condition
* Fluency in the test language with excellent proficiency, as appropriate to perform speech testing
* Functional auditory nerve
* General health condition, psychological and emotional condition deemed compatible with the treatment and tests performed in this study
* Pre-operative assessment according to the local professional standards
* Candidate is highly motivated and has realistic expectations about the expected benefit of the implant and shall understand the importance of returning to the implant centre for regular speech processor programming, assessment sessions and training
* Realistic expectations, as deemed appropriate by the implanting surgeon/implant board
* Evidence of up-to-date vaccinations against meningitis, as per recommendations by the applicable national body
* Signed and dated informed consent before the start of any study-specific procedure

Exclusion Criteria:

* Lack of compliance with any inclusion criterion
* Previously having received an implant on the location chosen for placing the cochlear implant
* Having received a hearing implant from another manufacturer than MED-EL on the contralateral ear
* Pre-existing condition known to necessitate MRI scans after implantation of the Mi2000 TICI
* Women being pregnant or nursing
* Women of childbearing age not reporting to use effective contraception
* The individual is known to be intolerant of the materials used in the implant or other required accessories including medical grade silicone, parylene C, titanium, platinum iridium, platinum, stainless chromate steel, thermoplastic elastomere (TPE-S), thermoplastic elastomere (SEBS), mixture of polycarbonate and acrylonitrile-butadiene-styrol polymer (PC/ABS), polyamide, liquid crystal polymer, silicone and polyurethane-coated silicone rubber)
* Absence of cochlear development
* The cause of deafness is non-functionality of the auditory nerve and/or the upper auditory pathway
* Medical contra-indications to middle ear and/or inner ear surgery, and/or anaesthesia
* External or middle ear infections are present
* The tympanic membrane is perforated in the ear to be implanted
* Anatomic abnormalities are present that would prevent appropriate placement of the stimulator housing in the bone of the skull, or prevent placement of the chosen electrode array into the cochlea (including ossification of the cochlea)
* The psychological status of the individual is unstable
* The individual has unrealistic expectations
* Acute cholesteatoma
* History of vestibular schwannoma
* Unstable Meniere's disease
* Auditory Neuropathy
* Epilepsy not responding to treatment
* Permanent inability and/or unwillingness to participation in post-operative care and rehabilitation
* Known intellectual disability and/or psychological diseases
* Participation in other pharmacological clinical trials within four weeks prior to enrolment
* Anything that, in the opinion of the Investigator, would place the subject at increased risk; preclude the subject's full compliance with or completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Word Test in Quiet | Pre-op to 6 months after first fitting
  Word test in quiet

SECONDARY OUTCOMES:
Health Utility Index Mark 3 (HUI3) | Pre-op to 6 months after first fitting
  Generic Quality of Life
Nijmegen Cochlear Implant Questionnaire (NCIQ) | Pre-op to 6 months after first fitting
  Disease specific Quality of Life

OTHER OUTCOMES:
Word test in quiet | through study completion, an average of 6 months after first fitting
  Word test in quiet
Sentence Test in Noise | 3- and 6-months after first fitting
  Oldenburg Matrix Test
Speech, Spatial, Quality of Hearing (SSQ12) | through study completion, an average of 6 months after first fitting
  Speech, Spatial and Quality of hearing scale
Hearing Implant Sound Quality Index (HISQUI) | through study completion, an average of 6 months after first fitting
  Sound quality questionnaire
Audiograms | through study completion, an average of 6 months after first fitting
  Audiograms

CONTACTS AND LOCATIONS:
Overall Officials: Florian Schwarze, PhD, Study Director — MED-EL Elektromedizinische Geräte GesmbH
Locations (6):
- AKH Wien, Vienna, Austria
- Belgium (2):
  - UZA Antwerpen, Antwerp
  - CHU Liège, Liège
- Germany (2):
  - LMU Munich, München, Bavaria
  - UKW Würzburg, Würzburg, Bavaria
- The Institute of Physiology and Pathology of Hearing, Nadarzyn, Poland

IPD SHARING:
Plan to Share IPD: No